CLINICAL TRIAL: NCT01854216
Title: Parallel Group Trial to Evaluate the Pharmacokinetics and Safety/Tolerability of Repeated Dose Treatment With Rotigotine Continuous Delivery System (5 cm^2/2.25 mg, 10 cm^2/4.5 mg, 20 cm^2/9 mg) in Japanese and Caucasian Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetics, Safety, Tolerability of Repeated Dose Transdermal Rotigotine in Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SP0718
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: Rotigotine; Neupro; Japanese; Caucasian; Male; Female; Single dose; Pharmacokinetics
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine in Japanese subjects (Experimental): Repeated-Dose application of 1,2, and 4 mg / 24 hours Rotigotine in healthy Japanese subjects; Transdermal patch over 24 hours
  Interventions: Drug: Rotigotine transdermal patch 1mg / 24 hours; Drug: Rotigotine transdermal patch 2 mg / 24 hours; Drug: Rotigotine transdermal patch 4 mg / 24 hours
- Rotigotine in Caucasian subjects (Experimental): Multiple-Dose application of 1, 2, and 4 mg / 24 hours Rotigotine in healthy Caucasian subjects; Transdermal patch over 24 hours
  Interventions: Drug: Rotigotine transdermal patch 1mg / 24 hours; Drug: Rotigotine transdermal patch 2 mg / 24 hours; Drug: Rotigotine transdermal patch 4 mg / 24 hours

INTERVENTIONS:
Drug: Rotigotine transdermal patch 1mg / 24 hours — Rotigotine transdermal patch, repeated dose application over 24 hours; 1 mg / 24 hours
  Other Names: Neupro
Drug: Rotigotine transdermal patch 2 mg / 24 hours — Rotigotine transdermal patch, repeated dose application over 24 hours; 2 mg / 24 hours
  Other Names: Neupro
Drug: Rotigotine transdermal patch 4 mg / 24 hours — Rotigotine transdermal patch, repeated dose application over 24 hours; 4 mg / 24 hours
  Other Names: Neupro

SUMMARY:
To investigate the repeated dose Pharmacokinetics (PK) of transdermally delivered Rotigotine in Japanese and Caucasian female and male healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy according to assessments done at eligibility assessment (medical history, physical examination, blood pressure, heart rate, ECG, hematology, clinical chemistry, urinalysis)
* Subject is of normal body-weight as determined by a body mass index ranging between 18 to 28 kg/m²
* Subject is Japanese or Caucasian. Japanese subjects are born in Japan and left Japan not more than 10 years ago. Both parents of the Japanese subjects are 100 % Japanese

Exclusion Criteria:

* Subjects (females) without medically adequate contraception or on lactation or pregnant women. Subjects with oral contraception or hormone replacement within 4 weeks prior to eligibility assessment
* Subject has a history of chronic alcohol or drug abuse
* Subject has a consumption of more than 20 g of alcohol/day (amount corresponds to 0.5 l of beer/day or 0.25 l of wine/day or 3 glasses (à 2 cl) of liquor/day)
* Subject has a clinically relevant allergy
* Subject has a known or suspected drug hypersensitivity in particular, to any component of the trial medication
* Subject has any clinically significant abnormality in physical examination
* Subject has a heart rate at rest less than 50 beats per minute (bpm) or more than 100 bpm
* Subject has systolic blood pressure lower than 100 mmHg or higher than 145 mmHg or diastolic blood pressure higher than 95 mmHg or lower than 60 mmHg
* Subject has an atopic or eczematous dermatitis and/or an active skin disease or skin tumors
* Subject has a history of significant skin hypersensitivity to adhesives or other transdermal products or recent unresolved contact dermatitis

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2002-12; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of unconjugated Rotigotine in steady-state within one dosing interval (AUCtau,ss) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Area under the concentration-time curve of unconjugated Rotigotine in steady-state within one dosing interval normalized by Body Weight [AUCtau,ss,norm(BW)] | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Maximum concentration of unconjugated Rotigotine in plasma at steady-state (Cmax,ss) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Maximum concentration of unconjugated Rotigotine in plasma at steady-state normalized by Body Weight [Cmax,ss,norm(BW)] | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Maximum concentration of unconjugated Rotigotine in plasma at steady-state normalized by apparent dose [Cmax,ss,norm(appd)] | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Maximum concentration of unconjugated Rotigotine in plasma at steady-state normalized by Body Weight and apparent dose [Cmax,ss,norm(BW,appd)] | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Area under the concentration-time curve of total Rotigotine in steady-state within one dosing interval (AUCtau,ss) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Area under the concentration-time curve of total Rotigotine in steady-state within one dosing interval normalized by Body Weight [AUCtau,ss,norm(BW)] | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Maximum concentration of total Rotigotine in plasma at steady-state (Cmax,ss) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Maximum concentration of total Rotigotine in plasma at steady-state normalized by Body Weight [Cmax,ss,norm(BW)] | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Maximum concentration of total Rotigotine in plasma at steady-state normalized by apparent dose [Cmax,ss,norm(appd)] | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Maximum concentration of total Rotigotine in plasma at steady-state normalized by Body Weight and apparent dose [Cmax,ss,norm(BW,appd)] | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours

SECONDARY OUTCOMES:
Terminal half-life (t1/2) of unconjugated Rotigotine in steady-state | Blood sampling at 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours
Time of maximum concentration (tmax) of unconjugated Rotigotine in steady-state (tmax,ss) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Apparent total body clearance of unconjugated Rotigotine normalized by Body Weight (CL/f/BW) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Apparent volume of distribution of unconjugated Rotigotine normalized by Body Weight (Vz/f/BW) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours
Terminal half-life (t1/2) of total Rotigotine in steady-state | Blood sampling at 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours
Time of maximum concentration (tmax) of total Rotigotine in steady-state (tmax,ss) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Apparent total body clearance of total Rotigotine normalized by Body Weight (CL/f/BW) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Apparent volume of distribution of total Rotigotine normalized by Body Weight (Vz/f/BW) | Blood sampling at 0 hours (predose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 1, Neuss, Germany

REFERENCES:
- [Derived] Cawello W, Kim SR, Braun M, Elshoff JP, Masahiro T, Ikeda J, Funaki T. Pharmacokinetics, safety, and tolerability of rotigotine transdermal system in healthy Japanese and Caucasian subjects following multiple-dose administration. Eur J Drug Metab Pharmacokinet. 2016 Aug;41(4):353-62. doi: 10.1007/s13318-015-0273-6. Epub 2015 Mar 13. PMID 25773763